CLINICAL TRIAL: NCT03996655
Title: Sugammadex Versus Neostigmine in Pediatric Day-case Cancer Surgery
Brief Title: Different Reversal Agents in Pediatric Day-case Cancer Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Amani Gaber Mohamed,MSc, Senior registra, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Reversal agents in pediatrics
Record Dates: First submitted 2019-06-18; First posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Post-operative Residual Curarization
MeSH Terms: interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group S (Experimental): Sugammadex for reversal of steroidal neuromuscular blockers, intravenous injection ,2mg/kg
  Interventions: Drug: Sugammadex Injection [Bridion]
- Group N (Active Comparator): Reversal of neuromuscular blockers, iv injection, 0.05 mg/kg
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: Sugammadex Injection [Bridion] — Reversal of neuromuscular blockers
  Arms: Group S
Drug: Neostigmine — Reversal of neuromuscular blockers
  Arms: Group N

SUMMARY:
The aim of this study was to compare the efficacy of sugammadex and neostigmine on

reversing neuromuscular blockers in pediatric patients undergoing outpatient surgical

procedures.

DETAILED DESCRIPTION:
Postoperative residual curarization (PORC)" a residual duration of action of muscle relaxants beyond the end of the operation" in postoperative patients is a succession of the presence of blocked nicotinic receptors. Even in observationally asymptomatic patients, 60-70% of these receptors can be still blocked. PORC can cause delayed recovery, hypoxia, metabolic derangement and rarely death. Cholinesterase inhibitors are traditionally used for reversal of neuromuscular blockade (NMB). Among these agents neostigmine is the most potent and selective one. Cholinesterase inhibitors have multisystemic side effects. Since these agents are not selective to nicotinic receptors and also stimulate the muscarinic system, there can be quite a few serious adverse effects as follows: Bradycardia, QT lengthening, bronchoconstriction, hypersalivation and increased motility. To avoid these effects, concomitant anticholinergic agents, such as atropine or glycopyrolate, are administered to the patient. The incidence of PORC is still high with the prevalence of a train-of-four (TOF) ratio of less than 0.9 found in the postoperative recovery unit. Recent studies have been able to link even low levels of residual paralysis (TOF ratio <0.9) with significant impairment of pharyngeal muscle function, hypoxic ventilatory drive and decreased respiratory function in the immediate postoperative period.

Despite the knowledge of such side effects, and despite the introduction of various new neuromuscular blocking agents (NMBA) such as rocuronium or mivacurium over the last 15 years, no significant reduction in the incidence of residual neuromuscular blockade has so far been observable.

Today, sugammadex is an alternative to the decurarization procedure, which was traditionally executed with cholinesterase inhibitors. Sugammadex a γ-cyclodextrin with a high affinity to rocuronium and other aminosteroidal NMBA that allows the rapid and complete reversal of especially rocuronium-induced neuromuscular blockade, has raised hopes to overcome the problem of residual neuromuscular blockade. Sugammadex is proved to be a safe and superior agent in NMB reversal compared to neostigmine in adults.

PORC and the muscarinic side effects are not anticipated when using sugammadex,.

Also, due to its pharmacodynamic profile, sugammadex, in combination with rocuronium, have the potential to displace succinylcholine as the "gold standard" muscle relaxant for rapid sequence induction.

The rudimentary neuromuscular junction, the variability of fibrin fibers, the differences in drug distribution and body volume in children change their neuromuscular conduction. These factors can cause prolonged recovery and increased risk of PORC. However, there is few studies in the literature concerning sugammadex administration in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥2 years and < 18 years.
* American society of anesthesiologists (ASA) status 1-3.
* patients undergoing outpatient procedures

Exclusion Criteria:

* Known drug hypersensitivity.-
* History of renal or hepatic failure.
* Diseases of the neuromuscular junction.
* history of malignant hyperthermia.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Recovery time | time from reversal administration until TOF ratio reaches0.9%, ranging from 1 to 2.5 minutes, measured withThe train-of-four (TOF) equipment working with the nerve-muscle acceleromyometry principle (TOF Draeger Medical Systems, Inc.16 Electronic Avenue,
  time from neostigmine or sugammadex administration until recovery of the TOF ratio to 0.9%

SECONDARY OUTCOMES:
extubation time | time from muscle relaxant administration until extubation,extubation will be performed based on clinical criteria extubation timeis estimated to range from 50 to 55 minutes
  time from neuromuscular blocker administration to extubation

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed MO Hegazy, MD, Study Director — Cairo University; Mohamed Ad Elramly, MD, Study Director — Cairo University

REFERENCES:
- [Background] Ammar AS, Mahmoud KM, Kasemy ZA. A comparison of sugammadex and neostigmine for reversal of rocuronium-induced neuromuscular blockade in children. Acta Anaesthesiol Scand. 2017 Apr;61(4):374-380. doi: 10.1111/aas.12868. Epub 2017 Feb 10. PMID 28185260
- [Background] Meretoja OA. Neuromuscular block and current treatment strategies for its reversal in children. Paediatr Anaesth. 2010 Jul;20(7):591-604. doi: 10.1111/j.1460-9592.2010.03335.x. PMID 20642658